CLINICAL TRIAL: NCT07244991
Title: Effect of MI Paste Plus™ on Streptococcus Mutans Counts and White Spot Lesions in Patients With Fixed Orthodontic Appliances: A Triple-Blind Clinical Trial
Brief Title: Effect of MI Paste Plus™ on Streptococcus Mutans and White Spot Lesions in Fixed Orthodontics
Acronym: MIPASTEORTHO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Beaty Dent (Other); Institute of Public Health, Albania (Other Government)
Responsible Party: Principal Investigator, Santiago Arias de Luxán, Professor of Orthodontics, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEEI25_585-Cardenal Herrera
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dental Caries; Streptococcus Mutans; Tooth Demineralization; Orthodontic Appliances, Fixed
Keywords: MI Paste Plus; Remineralization; Streptococcus mutans; White Spot Lesions; Fixed Orthodontic Appliances; Quantitative Light-Induced Fluorescence; Randomized Controlled Trial; Triple-Blind Study; Albania; CEU Cardenal Herrera University
MeSH Terms: conditions — Dental Caries; Tooth Demineralization | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups: the experimental group using MI Paste Plus (containing CPP-ACP and fluoride) and the control group using a bioadhesive placebo gel without active ingredients. Both groups will be followed concurrently for three months under identical clinical and microbiological evaluation schedules. The study follows a triple-blind design (participant, investigator, and outcome assessor) with stratified randomization by age, oral-hygiene risk, and type of orthodontic appliance.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is conducted under a triple-blind design. Participants, investigators, and outcome assessors remain unaware of group assignments. Both MI Paste Plus and placebo gels are identical in packaging, texture, and color and are supplied in coded opaque containers prepared by a dental hygienist not involved in patient evaluation or data analysis. The randomization code will be kept sealed until the completion of data collection and statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: MI Paste Plus (Experimental): Participants assigned to the experimental group will apply MI Paste Plus (GC Corporation, Japan) once daily at night after toothbrushing for three months. The product contains casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) and 0.20% sodium fluoride (≈900 ppm F-). Application is performed using a clean finger or applicator, avoiding eating, drinking, or rinsing for at least 30 minutes afterward. The goal is to evaluate the preventive effect of MI Paste Plus on Streptococcus mutans levels and enamel white-spot lesions during fixed orthodontic treatment.
  Interventions: Other: MI Paste Plus (CPP-ACP with Sodium Fluoride)
- Placebo Comparator: Bioadhesive Gel without Active Ingredients (Placebo Comparator): Participants in the control group will use an identical-appearing bioadhesive oral gel without active ingredients, applied once daily at night after toothbrushing for three months. The gel has the same texture, color, and packaging as MI Paste Plus and serves as the placebo control. Application instructions are identical to those of the experimental group.
  Interventions: Other: Bioadhesive Oral Gel (Placebo)

INTERVENTIONS:
Other: MI Paste Plus (CPP-ACP with Sodium Fluoride) — Participants in the experimental arm will apply MI Paste Plus once daily at night after toothbrushing for three months. MI Paste Plus is a water-based topical dental cream containing 10% casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) and 0.20% sodium fluoride (900 ppm F-). The product is applied using a clean finger or applicator and left undisturbed for at least 30 minutes. The intervention aims to reduce Streptococcus mutans counts and prevent enamel demineralization (white-spot lesions) during fixed orthodontic treatment.
  Arms: Experimental: MI Paste Plus
Other: Bioadhesive Oral Gel (Placebo) — Bioadhesive oral gel without active ingredients, identical in appearance to MI Paste Plus, applied once daily for three months under the same conditions to maintain blinding.
  Arms: Placebo Comparator: Bioadhesive Gel without Active Ingredients

SUMMARY:
Background This study is part of a doctoral research project at Universidad Cardenal Herrera CEU (Spain), directed by Prof. Santiago Arias de Luxán and conducted by doctoral candidate Shirli Kelmendi within the PhD program in Translational Medicine.

Fixed orthodontic appliances complicate oral hygiene by creating retention areas that favor bacterial colonization and alter microbial balance. These conditions increase plaque accumulation and Streptococcus mutans (S. mutans) proliferation in saliva and plaque. The frequent low-pH environment favors aciduric bacteria such as S. mutans and lactobacilli, promoting enamel demineralization and formation of white spot lesions (WSLs) or cavitations. WSLs appear as opaque white areas due to subsurface mineral loss, mainly in the gingival third of the crown. They may develop as early as one month after bracket placement, while in patients without appliances, progression occurs after at least six months. Increased S. mutans levels have been reported as early as six weeks after treatment start. Risk factors include poor brushing, lack of floss or rinse use, time since last cleaning, and presence of caries or lesions.

Intervention MI Paste Plus (GC, Japan) is a remineralizing cream with 0.20% sodium fluoride (900 ppm) and 10% CPP-ACP (RECALDENT™), providing calcium and phosphate stabilized by casein phosphopeptides. It has antibacterial and remineralizing effects, suitable during or after orthodontic treatment to prevent or reduce WSLs.

Objective To evaluate whether MI Paste Plus during fixed orthodontic treatment reduces S. mutans counts in saliva and/or WSL incidence.

Study Design A prospective, triple-blind, randomized clinical trial, approved by the Ethics Committee of the Ministry of Health of Albania and the Ethics Committee for Human Research of Universidad Cardenal Herrera CEU, Spain.

The study will include 200 patients (100 per group) from two orthodontic clinics in Tirana, Albania. Participants will be stratified by age, risk level, and appliance type, then randomized by third parties.

Outcome Measures Primary variables: S. mutans counts in saliva and number of WSLs after 3 months.

Standardized saliva collection, culturing, and bacterial quantification ensure consistency. Clinical assessments will be performed at 1 and 3 months using QRay Cam Pro (Inspektor Systems, Netherlands) for quantitative fluorescence and ICDAS for visual inspection.

Data will be analyzed using SPSS/R Commander software.

DETAILED DESCRIPTION:
Fixed orthodontic appliances are among the most common treatments in contemporary dentistry, yet they significantly modify the oral environment and create plaque-retentive areas that favor bacterial colonization. Brackets, ligatures, and auxiliary components increase the difficulty of oral hygiene and shift the ecological balance of the dental biofilm, favoring aciduric and acidogenic organisms such as Streptococcus mutans (S. mutans). Repeated exposure of dental plaque to a low pH inhibits acid-sensitive species and promotes S. mutans and lactobacilli, whose metabolic activity produces lactic acid and leads to enamel demineralization. Clinically, this presents as white-spot lesions (WSLs), the earliest visible stage of dental caries. Such lesions may appear within one month of appliance placement, whereas comparable demineralization in patients without orthodontic devices usually requires six months or longer. WSLs compromise esthetics and tooth integrity and may persist after orthodontic treatment ends, making early prevention essential.

Fluoride remains the most validated anti-caries agent, and the combination of fluoride with casein phosphopeptide-amorphous calcium phosphate (CPP-ACP) enhances remineralization by maintaining calcium and phosphate in bioavailable form. MI Paste Plus (GC Corporation, Japan) is a topical cream containing 10% CPP-ACP and 0.20% sodium fluoride (≈900 ppm F-), which releases calcium, phosphate, and fluoride ions that penetrate enamel, support remineralization, and inhibit bacterial ATPase activity. Although promising, further rigorously designed, adequately powered randomized clinical trials are needed to determine whether MI Paste Plus reduces salivary S. mutans levels and prevents WSLs during early orthodontic treatment. This doctoral research project aims to fill this gap.

The main objectives are to determine whether daily use of MI Paste Plus alters salivary S. mutans counts after one and three months of fixed orthodontic treatment and whether it prevents or reduces the incidence and severity of WSLs during the same period. Secondary objectives include assessing the relationship between oral hygiene risk status and baseline S. mutans levels or WSL prevalence, and examining whether age, hygiene risk, or appliance type modifies these outcomes. Null hypotheses state that MI Paste Plus does not significantly affect S. mutans levels or WSL development and that age, hygiene level, and appliance type do not modify these results.

This prospective, triple-blind, parallel-group randomized controlled clinical trial will take place in two private orthodontic polyclinics in Tirana, Albania. Ethical approval has been obtained from the Ministry of Health of Albania (Report No. 66/18, April 4, 2024) and from Universidad Cardenal Herrera CEU (May 12, 2025). All procedures comply with the Declaration of Helsinki, Good Clinical Practice, GDPR, the Spanish LOPD, and Albanian data protection law.

A sample of 200 patients (100 per group) will provide >90% power at α = 0.05 to detect moderate between-group differences, allowing for 10% attrition. Eligible participants will be 5-45 years old, beginning fixed orthodontic treatment, able to comply with procedures, and providing informed consent or assent. Exclusion criteria include systemic conditions affecting salivary flow, antimicrobial use within four weeks, allergies to milk proteins or fluoride, extensive restorations preventing enamel evaluation, or inability to attend follow-ups.

Participants will be stratified by age (≤15 or >15 years), oral hygiene risk (good or poor), and appliance type, then randomized 1:1 using a computer-generated list prepared by the study statistician. Allocation concealment will use sealed opaque envelopes and coded containers prepared by an independent hygienist. Test and placebo gels are identical in appearance, texture, and packaging. Participants, clinical evaluators, and microbiologists will remain blinded until data lock.

The test group will apply MI Paste Plus nightly for three months after toothbrushing. The control group will apply an inactive bioadhesive gel in the same manner. All participants will continue brushing with fluoridated toothpaste. Adherence will be monitored by daily logs and weighing returned containers.

Assessments occur at baseline (T0), one month (T1 ± 7 days), and three months (T2 ± 14 days). Clinical evaluation of WSLs will be performed using ICDAS. Teeth will be cleaned and dried for approximately five seconds using compressed air to enhance visibility of early changes. A dental operating light, mirror, and blunt probe will be used to classify surfaces from 0 to 6. Surfaces with ICDAS 0 at baseline will be considered sound; those that become ICDAS 1 or 2 at follow-up will be classified as new WSLs. For surfaces with ICDAS 1-2 at baseline, changes over time will indicate progression, stability, or improvement.

Quantitative Light-Induced Fluorescence (QLF™) imaging using the Q-Ray Cam Pro (Inspektor Systems, Netherlands) will complement ICDAS. QLF detects demineralized enamel as dark areas due to fluorescence loss and identifies porphyrin-producing bacterial activity as red/orange fluorescence. White-spot analysis will be performed in the software by activating the White Spot Analysis wizard. The system automatically generates several quantitative parameters, including ΔF (% fluorescence loss), ΔF max, ΔF Average, lesion area (WS Area), and porphyrin fluorescence metrics (ΔR, ΔR max, ΔR area). Although all parameters support clinical interpretation, only ΔF (%) will serve as a registered outcome measure. Negative ΔF values indicate demineralization, while changes in ΔF, WS Area, and ΔR patterns over time allow detection of new lesions and assessment of whether existing lesions progress, stabilize, or remineralize.

Stimulated saliva samples will be collected at least two hours after eating or brushing, refrigerated at 4 °C, and processed within 24 hours. Serial dilutions will be plated on TYCSB medium and incubated anaerobically for 72 hours. Colonies will be subcultured, identified using API 20 Strep, and quantified using standard CFU calculations. Two microbiologists will count plates independently.

Primary outcomes include salivary S. mutans counts and the presence, number, and severity of WSLs based on ICDAS and QLF ΔF values at T1 and T2. Secondary outcomes include plaque index, DMFT/DMFS, and associations with age, hygiene risk, and appliance type. Analyses will follow the intention-to-treat principle. Appropriate parametric or nonparametric tests and mixed-effects models will be used. Missing data will be addressed using multiple imputation.

All data will be recorded on paper CRFs and double-entered into a secure database. Calibration of ICDAS scoring, QLF imaging, and microbiological procedures will occur every six months. Adverse events are expected to be minor. Participants may withdraw at any time. Data confidentiality will follow GDPR, LOPD, and Albanian privacy regulations.

The preparatory phase is 90% complete, including protocol finalization, equipment procurement, staff training, and validation of all clinical and laboratory procedures. Recruitment will occur from November 2025 to June 2027, followed by analysis and dissemination. Results will be submitted to peer-reviewed journals in orthodontics, preventive dentistry, and microbiology, and presented at major conferences. A plain-language summary will be provided to participants, and anonymized datasets may be shared upon request under data-sharing agreements.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 45 years.
* Indication for fixed orthodontic treatment, either with fixed auxiliary appliances (including orthopedic devices) or brackets with or without auxiliary components.
* General good health with no systemic diseases affecting oral health.

Exclusion Criteria:

* Advanced white-spot lesions with untreated dentin involvement.
* Presence of active untreated dental caries at baseline.
* Antibiotic therapy within the previous two months.
* Previous diagnosis of molar-incisor hypomineralization (MIH).
* History of immunosuppression.
* Iron-deficiency anemia or other clinically relevant hematological disorders.
* Parafunctional habits such as lip sucking or finger sucking.
* Use of any type of dental prosthesis.
* Smoking or tobacco use.
* Documented allergy to nickel.
* Requirement for orthodontic treatment using removable appliances or clear aligners.

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in salivary Streptococcus mutans count (log₁₀ CFU/mL) | Baseline, 1 month, 3 months
  Stimulated saliva will be collected after ≥2 hours of fasting and oral hygiene abstention, using sterile insulin syringes to obtain 2-3 mL directly from the floor of the mouth. Samples will be refrigerated (4 °C, ≤24h), serially diluted in saline, and 1 µL plated onto TYCSB selective agar for anaerobic incubation at 37 °C for 72 hours. Colonies will be identified morphologically and confirmed with API Strep 20. S. mutans levels (CFU/mL) will be calculated from colony counts and dilution factors and expressed as log₁₀ CFU/mL. The outcome is the change in S. mutans from baseline to 1 and 3 months.

SECONDARY OUTCOMES:
Incidence of new white-spot enamel lesions detected by ICDAS | Baseline, 1 month, 3 months
  White-spot enamel lesions will be assessed using the International Caries Detection and Assessment System (ICDAS). Teeth are cleaned, dried for 5 seconds with compressed air, and examined using a dental operating light, mirror, and blunt probe.
  A tooth surface will be considered sound at baseline if it has ICDAS score 0. A new white-spot lesion is defined as a surface that was ICDAS 0 at baseline and presents ICDAS 1 or 2 at the 3-month examination.
  The outcome is the proportion of participants who develop at least one new ICDAS-detected white-spot lesion during the 3-month follow-up.
Change in ΔF (%) of white-spot lesions measured by QLF™ | Baseline, 1 month, 3 months
  White-spot enamel lesions will be evaluated using Quantitative Light-Induced Fluorescence (QLF™) with the QRay Cam Pro (Inspektor Systems, Netherlands). Dark areas in QLF images represent enamel demineralization (fluorescence loss), while areas with bacterial porphyrins show red/orange fluorescence.
  White-spot analysis will be performed using the QLF software ("White Spot Analysis" tab). After selecting the lesion location, the white-spot wizard will generate quantitative parameters.
  The primary fluorescence parameter reported for this study will be ΔF (%), which represents the percentage loss of fluorescence relative to sound enamel and correlates with lesion depth.
  This outcome will capture the development of new white-spot lesions (new negative ΔF values on previously sound surfaces) and the progression or improvement of pre-existing lesions over the 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Arias de Luxán, DMD, PhD, Principal Investigator — Universidad CEU Cardenal Herrera - Facultad de Ciencias de la Salud
Locations (2):
- Albania (2):
  - Beaty Dent, Tirana, Albania
  - Happy Dent, Tirana, Albania

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available to protect patient privacy, but de-identified data may be provided by the corresponding author upon reasonable request after publication.

REFERENCES:
- [Background] Wan AK, Seow WK, Walsh LJ, Bird PS. Comparison of five selective media for the growth and enumeration of Streptococcus mutans. Aust Dent J. 2002 Mar;47(1):21-6. doi: 10.1111/j.1834-7819.2002.tb00298.x. PMID 12035953
- [Background] Maret D, Marchal-Sixou C, Vergnes JN, Hamel O, Georgelin-Gurgel M, Van Der Sluis L, Sixou M. Effect of fixed orthodontic appliances on salivary microbial parameters at 6 months: a controlled observational study. J Appl Oral Sci. 2014 Jan-Feb;22(1):38-43. doi: 10.1590/1678-775720130318. PMID 24626247
- [Background] Robertson MA, Kau CH, English JD, Lee RP, Powers J, Nguyen JT. MI Paste Plus to prevent demineralization in orthodontic patients: a prospective randomized controlled trial. Am J Orthod Dentofacial Orthop. 2011 Nov;140(5):660-8. doi: 10.1016/j.ajodo.2010.10.025. PMID 22051486
- See also: Official website of Universidad Cardenal Herrera CEU, the academic institution overseeing the doctoral research project. — https://www.uchceu.es/en